CLINICAL TRIAL: NCT06919588
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effects of Comedy Therapy on Anxiety and Vital Signs in Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan7
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant; Complications; Stress; Care Acceptor, Health
Keywords: stress; vital signs; pre-operative; liver; transplant; comedy films
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pretestpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comedy therapy (Experimental): Before transplant surgery, a patient introduction form and a state anxiety scale will be applied as a pre-test, and vital signs will be checked. Patients will be shown 10-minute Turkish comedy films prepared by researchers before transplant surgery. After the intervention, vital signs will be checked as a post-test, and a state anxiety scale will be applied. While patients are shown the comedy films, a quiet and calm environment will be provided in the patient room.
  Interventions: Behavioral: comedy therapy
- standard of care (No Intervention): Before transplant surgery, a patient introduction form and a state anxiety scale will be applied as a pre-test, and vital signs will be checked. No intervention will be made to the control group patients outside of the clinical protocol. After a certain waiting period (average of 30 minutes), the patients' vital signs will be checked and the state anxiety scale will be applied again.

INTERVENTIONS:
Behavioral: comedy therapy — Before the transplant surgery, the patients were shown 10-minute Turkish comedy films prepared by the researchers.
  Arms: comedy therapy

SUMMARY:
This study was conducted to investigate the effects of watching excerpts from classical Turkish comedy films on pre-transplant anxiety levels and vital signs in liver transplant recipients.

H1-0: Watching classical Turkish comedy films has no effect on preoperative anxiety in liver transplant recipients.

H1-1: Watching classical Turkish comedy films reduces preoperative anxiety in liver transplant recipients.

H2-0: Watching classical Turkish comedy films has no effect on preoperative vital signs in liver transplant recipients.

H2-1: Watching classical Turkish comedy films has a positive effect on preoperative vital signs in liver transplant recipients.

DETAILED DESCRIPTION:
Intervention Group:

A patient introduction form and a state anxiety scale will be applied as a pre-test before transplant surgery, and vital signs will be checked. Patients will be shown 10-minute Turkish comedy films prepared by researchers before transplant surgery. After the intervention, vital signs will be checked as a post-test and a state anxiety scale will be applied. A quiet and calm environment will be provided in the patient room while patients are shown the comedy films.

Control Group:

A patient introduction form and a state anxiety scale will be applied as a pre-test before transplant surgery, and vital signs will be checked. No intervention will be made to the control group patients outside of the clinical protocol. After a certain waiting period (average of 30 minutes), the patients' vital signs will be checked and the state anxiety scale will be applied again.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Being a liver transplant recipient,
* Data obtained before transplantation,
* Not having any visual or auditory problems.

Exclusion Criteria:

* Being under 18 years of age,
* Having any visual/auditory problems,
* Not accepting to participate in the study/wanting to leave,
* Not providing hemodynamic instability (sudden change in vital signs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
anxiety level | Between April and August.
  The anxiety levels of patients will be measured using the "State and Trait Anxiety Scale".
  State and Trait Anxiety Scale; consists of two scales. Each scale has 20 questions. Scoring is between 1-4. Each scale score varies between 20-80 points. A high scale score indicates high anxiety. A low scale score indicates low anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin Okutan, Dr., Principal Investigator — Study Principal Investigator Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)